CLINICAL TRIAL: NCT07292870
Title: Evaluation of the Addition of Different Biologicals in the Surgical Treatment of Periodontal Intra-Bony Defects: A Randomised Controlled Clinical Trial.
Brief Title: Biologicals in Management of Intra-Bony Defects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S69198
Record Dates: First submitted 2025-11-18; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-10

CONDITIONS: Intra-bony Pockets; Periodontitis
Keywords: Intra-bony defects; periodontitis; minimally invasive surgery; biologicals; L-PRF; Hyaluronic acid; enamel matrix derivative; leukocyte- and platelet-rich fibrin
MeSH Terms: conditions — Periodontitis | interventions — enamel matrix proteins; Leukocyte Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Bio-Oss® collagen + Emdogain® (Placebo Comparator): minimally invasive surgery + Bio-Oss® collagen + Emdogain® (MIS + BO + Enamel Matrix Derivative)
  Interventions: Procedure: Minimally invasive surgical treatment of the intra-bony defects; Procedure: Use of the xenograft Bio-Oss® Collagen during the surgery; Procedure: Use of enamel matrix derivative (Emdogain®)
- Bio-Oss® collagen + REGENFAST® (Active Comparator): minimally invasive surgery + Bio-Oss® collagen + REGENFAST® (MIS + BO + hyaluronic acid)
  Interventions: Procedure: Minimally invasive surgical treatment of the intra-bony defects; Procedure: Use of the xenograft Bio-Oss® Collagen during the surgery; Procedure: Use of hyaluronic acid (REGENFAST®)
- Bio-Oss® collagen + L-PRF (Active Comparator): minimally invasive surgery + Bio-Oss® collagen + L-PRF (MIS + BO + Leucocyte -Platelet Rich Fibrin)
  Interventions: Procedure: Minimally invasive surgical treatment of the intra-bony defects; Procedure: Use of the xenograft Bio-Oss® Collagen during the surgery; Procedure: use of the blood derivative L-PRF (leukocyte and platelet rich fibrin)
- L-PRF (Active Comparator): minimally invasive surgery + L-PRF (MIS + Leucocyte-Platelet Rich Fibrin)
  Interventions: Procedure: Minimally invasive surgical treatment of the intra-bony defects; Procedure: use of the blood derivative L-PRF (leukocyte and platelet rich fibrin)

INTERVENTIONS:
Procedure: Minimally invasive surgical treatment of the intra-bony defects — A surgical procedure is performed under local anaesthesia in which one of the biomaterials will be used to fill the intra-bony defect.
Procedure: Use of the xenograft Bio-Oss® Collagen during the surgery — The clinician will use Bio-Oss® Collagen as adjuvant in the surgical treatment of the intra-bony defects in conjunction with minimally invasive surgery
  Arms: Bio-Oss® collagen + Emdogain®; Bio-Oss® collagen + L-PRF; Bio-Oss® collagen + REGENFAST®
Procedure: Use of enamel matrix derivative (Emdogain®) — The clinician will use Enamel matrix derivative (Emdogain®) as adjuvant in the surgical treatment of the intra-bony defects in conjunction with minimally invasive surgery.
  Arms: Bio-Oss® collagen + Emdogain®
Procedure: Use of hyaluronic acid (REGENFAST®) — The clinician will use hyaluronic acid (REGENFAST®) as adjuvant in the surgical treatment of the intra-bony defects in conjunction with minimally invasive surgery
  Arms: Bio-Oss® collagen + REGENFAST®
Procedure: use of the blood derivative L-PRF (leukocyte and platelet rich fibrin) — The clinician will use L-PRF as adjuvant in the surgical treatment of the intra-bony defects in conjunction with minimally invasive surgery.
  Arms: Bio-Oss® collagen + L-PRF; L-PRF

SUMMARY:
The aim is of this study is to evaluate and compare the effects (clinical and radiological) of different biomaterials on the repair of bone defects around the teeth. When participating in this study, persons will be scheduled for local surgical intervention of the gums. Under local anaesthesia, the gums will be opened minimally to gain insight into the underlying bone defect. After the bone defect has been made completely free of inflammation, they will be randomly assigned to one of the groups below and the biomaterials for this group will be used to fill the defect around your teeth. The different biomaterials are artificial bone + amelogenin; artificial bone + hyaluronic acid; artificial bone + blood preparation (L-PRF) or blood preparation alone.

Then the gums will be closed again with a suture and they will receive the necessary instructions regarding the procedure.

DETAILED DESCRIPTION:
The purpose of this study is to assess the clinical and radiological effectiveness of hyaluronic acid (REGENFAST®), enamel matrix derivative (Emdogain®), and platelet concentrates (L-PRF) in the surgical treatment (minimally invasive technique) of intra-bony defects in conjunction with minimally invasive surgery..

This is a non-inferiority study. The alternative hypothesis is that the use of hyaluronic acid or L-PRF obtained at least the same treatment outcome (seen as clinical attachment level gain) than the gold standard (use of enamel matrix derivatives).

2.2. Primary Endpoints

Post-operative changes in clinical attachment level (CAL):

* difference between the baseline and 6/12 months after the surgery
* measured in millimetres

2.3. Secondary Endpoints

Post-operative changes in probing pocket depth (PPD):

* difference between the baseline and 6/12 months after the surgery
* measured in millimetres

Post-operative changes in papilla height (preservation of soft tissues):

* difference between the baseline and 6/12 months after the surgery
* measured by means of a volumetric analysis based on intra-oral scan

Post-operative changes in intra-bony defect morphology:

* difference between the baseline and 6/12 months after the surgery
* periapical radiograph (parallel angle technique)
* defect resolution measured in millimetres
* bone fill measured in percentage

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
* At least 18 years of age at the time of signing the Informed Consent Form (ICF)
* American Society of Anesthesiology (ASA) score I or II
* Has already completed the non-surgical periodontal therapy with remaining local pockets of ≥ 6 mm14
* The intra-bony defect should be non-contained (2-wall defect)
* Clinical indication for surgical treatment of the intra-bony defect with minimally invasive approach in conjunction with biologicals

Exclusion Criteria:

* Under the age of 18 years
* Any disorder, which in the Investigator's opinion might jeopardise the participant's safety or compliance with the protocol
* Any prior or concomitant treatment(s) that might jeopardise the participant's safety or that would compromise the integrity of the Trial
* Participation in an interventional Trial with an investigational medicinal product (IMP) or device
* Known or suspected current malignancy
* History of chemotherapy
* History of radiation in the head and neck region
* History of other metabolic bone diseases
* Current or previous use of intravenous and oral bisphosphonates
* Haematological disorders
* Pregnancy / lactation
* Smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative changes in clinical attachment level (CAL) | 6/12 months after surgery
  difference between the baseline and 6/12 months after the surgery measured in mm

SECONDARY OUTCOMES:
Post-operative changes in probing pocket depth (PPD) | 6/12 months after the surgery
  difference between the baseline and 6/12 months after the surgery measured in mm
Post-operative changes in papilla height (preservation of soft tissues) | 6/12 months after the surgery
  difference between the baseline and 6/12 months after the surgery measured by means of a volumetric analysis based on intra-oral scan
Post-operative changes in intra-bony defect morphology | 6/12 months after the surgery
  difference between the baseline and 6/12 months after the surgery, via periapical radiograph (parallel angle technique); defect resolution measured in millimetres and bone fill measured in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Ana Castro, Professor, Principal Investigator — UZLeuven, department of Oral Health Sciences, Periodontology
Locations (1):
- UZLeuven, Campus St. Raphaël, Department Oral Health Sciences, Periodontology, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No